CLINICAL TRIAL: NCT00124982
Title: A Phase III, Multi-Center, Open Label Study to Evaluate the Efficacy, Tolerability and Safety of Abatacept (BMS-188667) in Subjects With Active Rheumatoid Arthritis on Background Non-Biologic DMARDs Who Have an Inadequate Response to Anti-TNF Therapy and Have Limited Therapeutic Options
Brief Title: Study of Abatacept (BMS-188667) in Subjects With Active Rheumatoid Arthritis on Background Non-biologic DMARDS (Disease Modifying Antirheumatic Drugs) Who Have an Inadequate Response to Anti-TNF Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-064
Record Dates: First submitted 2005-06-30; First posted 2005-07-29 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Therapeutics

ARMS (3):
- Open-label Abatacept (ABA)-Previous User (Experimental): In participants who have had an inadequate efficacy response or intolerance on previous TNF-antagonist therapy (off therapy for at least 2 months), open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
  Interventions: Drug: Abatacept; Drug: Non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)
- Open-label ABA-Current User (Experimental): In participants currently using Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
  Interventions: Drug: Abatacept; Drug: Non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD); Drug: Anti-Tumor Necrosing Factor (TNF) Therapy
- Long-term ABA (Experimental): Participants continued to receive the same 10 mg/kg weight-tiered dose of abatacept that they received in the initial short-term period.
  Interventions: Drug: Abatacept; Drug: Non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)

INTERVENTIONS:
Drug: Abatacept — IV solution, IV infusion, between 500mg and 1gram based on body weight, monthly, 6 months.
  Other Names: Orencia
Drug: Non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD) — During the study, subjects continued to receive 1 or more background non-biologic DMARDs (e.g. methotrexate, leflunomide) at the dose level(s) and regimen(s) administered at the time of abatacept treatment onset (Day 1).
Drug: Anti-Tumor Necrosing Factor (TNF) Therapy — Any of the anti-TNF therapies (Infliximab, Adalimumab, Etanercept, etc.)administered at the approved label dose for at least 3 months
  Arms: Open-label ABA-Current User

SUMMARY:
The purpose of this study is to summarize the safety and tolerability of abatacept during 6 months of combined treatment with one or more of the background non-biologic disease modifying anti-rheumatic drugs (DMARDs) approved for rheumatoid arthritis (RA) in subjects with active RA. Secondary objectives assessed the clinical efficacy of combination treatment, including disease activity, physical function, and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Completed double-blind portion of the IM101064 study.
* Rheumatoid arthritis (RA) for greater than 1 year from the time of initial diagnosis
* American College of Rheumatology (ACR) functional class I, II, III
* Subjects currently or previously received an anti-TNF therapy at an approved labeled dose for at least 3 months

Exclusion Criteria:

* Subjects with active vasculitis of a major organ system (except subcutaneous rheumatoid nodules)
* History of cancer within the last 5 years (other than non-melanoma skin cell cancers cured by local resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1286 (Actual)
Dates: Start 2005-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (148):
- United States (114):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Paradise Valley, Arizona
  - Local Institution, Peoria, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Long Beach, California
  - Local Institution, Palm Springs, California
  - Local Institution, Palo Alto, California
  - Local Institution, San Diego, California
  - Local Institution, Santa Monica, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Danbury, Connecticut
  - Local Institution, Hamden, Connecticut
  - Local Institution, Trumbull, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Aventura, Florida
  - Local Institution, Clearwater, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Largo, Florida
  - Local Institution, Sarasota, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Blue Ridge, Georgia
  - Local Institution, Macon, Georgia
  - Local Institution, Morton Grove, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Des Moines, Iowa
  - Local Institution, Kansas City, Kansas
  - Local Institution, Prairie Village, Kansas
  - Local Institution, Bowling Green, Kentucky
  - Local Institution, Louisville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Boston, Massachusetts
  - Local Institution, Peabody, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, East Lansing, Michigan
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Lansing, Michigan
  - Local Institution, Petockey, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Saint Paul, Minnesota
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Lebanon, New Hampshire
  - Local Institution, Nashua, New Hampshire
  - Local Institution, Cherry Hill, New Jersey
  - Local Institution, Dover, New Jersey
  - Local Institution, Manalapan, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Somerset, New Jersey
  - Local Institution, Teaneck, New Jersey
  - Local Institution, Voorhees Township, New Jersey
  - Local Institution, Albany, New York
  - Local Institution, Brooklyn, New York
  - Local Institution, Hewlett, New York
  - Local Institution, Lake Success, New York
  - Local Institution, Mineola, New York
  - Local Institution, New York, New York
  - Local Institution, Olean, New York
  - Local Institution, Orchard Park, New York
  - Local Institution, Rochester, New York
  - Local Institution, Schenectady, New York
  - Local Institution, Smithtown, New York
  - Local Institution, Syracuse, New York
  - Local Institution, Asheville, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Bismarck, North Dakota
  - Local Institution, Akron, Ohio
  - Local Institution, Beachwood, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Mayfield Village, Ohio
  - Local Institution, Youngstown, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Bala-Cynwyd, Pennsylvania
  - Local Institution, Bethlehem, Pennsylvania
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution, Duncansville, Pennsylvania
  - Local Institution, Erie, Pennsylvania
  - Local Institution, Meadville, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, West Reading, Pennsylvania
  - Local Institution, Wexford, Pennsylvania
  - Local Institution, Willow Grove, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Myrtle Beach, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Sioux Falls, South Dakota
  - Local Institution, Hixson, Tennessee
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Galveston, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Lubbock, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Sugarland, Texas
  - Local Institution, Burke, Virginia
  - Local Institution, Chesapeake, Virginia
  - Local Institution, Fairfax, Virginia
  - Local Institution, Salem, Virginia
  - Local Institution, Seattle, Washington
  - Local Institution, Vancouver, Washington
  - Local Institution, Glendale, Wisconsin
  - Local Institution, La Crosse, Wisconsin
  - Local Institution, Madison, Wisconsin
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Local Institution, Prague, Czechia
- France (10):
  - Local Institution, Boisguillaume
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Germany (5):
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Kiel
  - Local Institution, Leipzig
  - Local Institution, Tübingen
- Local Institution, Cork, Cork, Ireland
- Italy (3):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Torino
- Mexico (2):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Distrito Federal, Mexico City
- Spain (6):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Guipuzcoa
  - Local Institution, Madrid
  - Local Institution, Santander
  - Local Institution, Valencia
- United Kingdom (4):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Maidstone, Kent
  - Local Institution, Leeds, North Yorkshire

REFERENCES:
- [Background] Schiff M, Pritchard C, Huffstutter JE, Rodriguez-Valverde V, Durez P, Zhou X, Li T, Bahrt K, Kelly S, Le Bars M, Genovese MC. The 6-month safety and efficacy of abatacept in patients with rheumatoid arthritis who underwent a washout after anti-tumour necrosis factor therapy or were directly switched to abatacept: the ARRIVE trial. Ann Rheum Dis. 2009 Nov;68(11):1708-14. doi: 10.1136/ard.2008.099218. Epub 2008 Dec 15. PMID 19074911
- [Derived] Alten R, Burkhardt H, Feist E, Kruger K, Rech J, Rubbert-Roth A, Voll RE, Elbez Y, Rauch C. Abatacept used in combination with non-methotrexate disease-modifying antirheumatic drugs: a descriptive analysis of data from interventional trials and the real-world setting. Arthritis Res Ther. 2018 Jan 2;20(1):1. doi: 10.1186/s13075-017-1488-5. PMID 29329602
- [Derived] Vieira MC, Zwillich SH, Jansen JP, Smiechowski B, Spurden D, Wallenstein GV. Tofacitinib Versus Biologic Treatments in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors: Results From a Network Meta-analysis. Clin Ther. 2016 Dec;38(12):2628-2641.e5. doi: 10.1016/j.clinthera.2016.11.004. Epub 2016 Nov 24. PMID 27889300
- [Derived] Hassett AL, Li T, Buyske S, Savage SV, Gignac MA. The multi-faceted assessment of independence in patients with rheumatoid arthritis: preliminary validation from the ATTAIN study. Curr Med Res Opin. 2008 May;24(5):1443-53. doi: 10.1185/030079908x297376. Epub 2008 Apr 9. PMID 18402714
- [Derived] Genovese MC, Schiff M, Luggen M, Becker JC, Aranda R, Teng J, Li T, Schmidely N, Le Bars M, Dougados M. Efficacy and safety of the selective co-stimulation modulator abatacept following 2 years of treatment in patients with rheumatoid arthritis and an inadequate response to anti-tumour necrosis factor therapy. Ann Rheum Dis. 2008 Apr;67(4):547-54. doi: 10.1136/ard.2007.074773. Epub 2007 Oct 5. PMID 17921185

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1286 participants enrolled in this study, 240 were not treated.
Groups:
- Short Term (ST) Abatacept (ABA)-Previous User: In participants who had previously used Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
- ST-Current User: In participants currently using Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
Period: Short-term Period
Arm/Group | Short Term (ST) Abatacept (ABA)-Previous User | ST-Current User | Long-term ABA
Started | 449 | 597 | 0
Completed | 377 | 483 | 0
Not Completed | 72 | 114 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Adverse Event | 17 | 22 | 0
Not completed — Lack of Efficacy | 32 | 73 | 0
Not completed — Lost to Follow-up | 8 | 5 | 0
Not completed — Withdrawal of Consent | 7 | 9 | 0
Not completed — Poor/Non-compliance | 3 | 1 | 0
Not completed — No Longer Meets Study Criteria | 1 | 2 | 0
Not completed — Participant Decision | 1 | 0 | 0
Not completed — Participant Chose Own Doctor | 0 | 1 | 0
Not completed — Investigator Decision-No Specific AE | 1 | 0 | 0
Not completed — Participant Had Lymphopenia | 1 | 0 | 0
Period: Long-term Period
Arm/Group | Short Term (ST) Abatacept (ABA)-Previous User | ST-Current User | Long-term ABA
Started | 0 | 0 | 530 (A large number did not continue due to a rollover from study drug to commercially available drug.)
Completed | 0 | 0 | 441
Not Completed | 0 | 0 | 89
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 17
Not completed — Lack of Efficacy | 0 | 0 | 46
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 16
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Poor/Non-compliance | 0 | 0 | 2
Not completed — Administrative Reason by Sponsor | 0 | 0 | 1
Not completed — Neurologist Recommendation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ST Abatacept (ABA)-Previous User: In participants who had previously used Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
- ST ABA-Current User: In participants currently using Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
- Total: Total of all reporting groups
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User | Total
Number analyzed (Participants) | 449 | 597 | 1046
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.5) | 53.2 (12.3) | 54.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359 | 490 | 849
  Male | 90 | 107 | 197
Number of Tender Joints [Mean (Standard Deviation); unit: tender joints] — The mean number of tender joints was evaluated based on the number of tender joints in a standard 68 joint count.
  tender joints | 17.8 (5.9) | 17.8 (6.1) | 17.8 (6.0)
Number of Swollen Joints [Mean (Standard Deviation); unit: swollen joints] — The mean number of swollen joints was evaluated based on the number of swollen joints in a standard 66 joint count.
  swollen joints | 13.9 (5.6) | 13.5 (5.4) | 13.6 (5.5)
Physical Function, Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. HAQ-DI= sum of worst scores in each domain divided by the number of domains answered. HAQ-DI ranges from a minimum of 0 (no difficulty) to a maximum overall score of 3(unable to do).
  units on a scale | 1.7 (0.6) | 1.7 (0.6) | 1.7 (0.6)
hs-C-Reactive Protein (hs-CRP) Serum Levels [Mean (Standard Deviation); unit: mg/dL] — hs-CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of hs-CRP can be used to determine DAS28.
  mg/dL | 2.2 (3.0) | 2.1 (3.0) | 2.1 (3.0)
Disease Activity Score (DAS) 28 (Using CRP Levels) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, serum CRP level, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
  units on a scale | 6.2 (0.7) | 6.2 (0.7) | 6.2 (0.7)
Rheumatoid Factor (RF) Status [Number; unit: participants] — Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process.
  participants
    Negative | 138 | 215 | 353
    Positive | 292 | 349 | 641
    Data Not Available | 19 | 33 | 52

OUTCOME MEASURES:

1. Primary Outcome: Short-term Period: Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuations, AEs, Related AEs, or AEs Leading to Discontinuations
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with treatment.SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.Related AE/SAE=Certain,Probable,Possible,or Missing relationship to Drug
Time Frame: Days 1-169
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 449 | 597
participants
  Death | 1 | 1
  SAEs | 50 | 59
  Related SAEs | 10 | 16
  SAEs Leading to Discontinuation | 9 | 8
  AEs | 350 | 473
  Related AEs | 190 | 273
  AEs Leading to Discontinuation | 17 | 24

2. Primary Outcome: Short-term Period: Number of Participants With AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, and opportunistic infections; autoimmune disorders; neoplasms; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion).
Time Frame: Days 1-169
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 449 | 597
participants
  Infections (pre-specified) | 26 | 38
  Serious Infections (pre-specified) | 6 | 7
  Benign, malignant, and unspecified neoplasms | 8 | 7
  Autoimmune disorders (pre-specified) | 4 | 9
  Acute infusional AEs (pre-specified) | 20 | 37
  Peri-infusional AEs (pre-specified) | 57 | 99

3. Secondary Outcome: Short-term Period: Number of Participants With Clinically Meaningful Improvement (CMI) in Disease Activity Score (DAS 28), Low Disease Activity (LDAS), or Remission at Day 169
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
Time Frame: BL, Day 169
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 449 | 597
participants
  CMI | 267 | 320
  LDAS | 101 | 133
  Remission | 54 | 82

4. Primary Outcome: Short-term Period: Number of Participants With Hematology Laboratories Meeting Marked Abnormality (MA) Criteria
Description: Upper Normal Limit (ULN), Lower Normal Limit (LLN), Baseline (BL). Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use 0.5 * BL/<100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL/>ULN, or if BL>ULN then use >1.2 * BL/<LLN; neutrophils+bands: <1.0 * 10^3 c/uL; eosinophils: >0.750 * 10^3 c/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL.
Time Frame: Days 1-169
Population: Participants who received at least 1 infusion of abatacept during the short-term treatment period
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 429 | 581
participants
  Low HGB (n=429, n=581) | 2 | 3
  Low hematocrit (n=428, n=580) | 1 | 2
  Low erythrocytes (n=429, n=581) | 1 | 2
  Low PLT (n=424, n=578) | 1 | 1
  High PLT (n=424, n=578) | 0 | 0
  Low leukocytes (n=429, n=581) | 2 | 1
  High leukocytes (n=429, n=581) | 3 | 8
  Low neutrophils+bands (n=429, n=580) | 0 | 1
  High eosinophils (n=429, n=580) | 2 | 2
  High basophils (n=429, n=580) | 0 | 0
  High monocytes (n=429, n=580) | 1 | 0
  Low lymphocytes (n=429, n=580) | 30 | 27
  High lymphocytes (n=429, n=580) | 0 | 0

5. Primary Outcome: Short-term Period: Number of Participants With Liver and Kidney Function Laboratories Meeting MA Criteria
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; aspartate aminotransferase (AST): >3* ULN, or if BL>ULN then use >4* BL; alanine aminotransferase (ALT): >3* ULN, or if BL>ULN then use >4* BL; G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; Bilirubin: >2* ULN, or if BL>ULN then use >4* BL; blood urea nitrogen (BUN): >2* BL; creatinine: >1.5* BL
Time Frame: Days 1-169
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 428 | 583
participants
  High ALP (n=428, n=583) | 0 | 0
  High AST (n=426, n=583) | 1 | 2
  High ALT (n=426, n=583) | 2 | 1
  High GGT (n=427, n=583) | 1 | 5
  High bilirubin (n=426, n=583) | 1 | 1
  High BUN (n=428, n=583) | 3 | 8
  High creatinine (n=427, n=583) | 8 | 7

6. Primary Outcome: Short-term Period: Number of Participants With Electrolyte Laboratories Meeting MA Criteria
Description: Marked abnormality criteria:Sodium (Na): <0.95* LLN/ >1.05* ULN,or if BL<LLN then use 0.95* BL or >ULN,or if BL>ULN then use>1.05* BL or <LLN; potassium (K): <0.9* LLN/>1.1* ULN,or if BL<LLN then use 0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; chloride: <0.9* LLN/>1.1* ULN, or if BL<LLN then use 0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; calcium (Ca): <0.8* LLN/>1.2* ULN, or if BL<LLN then use 0.75* BL or >ULN, or if BL>ULN then use>1.25* BL or <LLN; phosphorous (P): <0.75* LLN/ >1.25* ULN, or if BL<LLN then use 0.67* BL or >ULN, or if BL>ULN then use>1.33* BL or <LLN
Time Frame: Days 1-169
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 428 | 583
participants
  Low Na (n=428, n=583) | 0 | 2
  High Na (n=428, n=583) | 0 | 0
  Low K (n=425, n=583) | 1 | 3
  High K (n=425, n=583) | 0 | 0
  Low chloride (n=428, n=583) | 0 | 0
  High chloride (n=428, n=583) | 0 | 0
  Low Ca (n=428, n=583) | 2 | 0
  High Ca (n=428, n=583) | 0 | 0
  Low P (n=426, n=583) | 1 | 0
  High P (n=426, n=583) | 3 | 1

7. Primary Outcome: Short-term Period: Number of Participants With Other Chemistry and Urinalysis Laboratories Meeting MA Criteria
Description: Marked abnormality criteria: serum glucose (Glu):<65 mg/dL/ >220 mg/dL; fasting serum Glu: <0.8* LLN/>1.5* ULN, or if BL<LLN then use 0.8* BL or >ULN, or if BL>ULN then use >2.0* BL or <LLN; total protein: <0.9* LLN/>1.1* ULN; albumin: <0.9* LLN,or if BL<LLN then use <0.75 BL; uric acid: >1.5* ULN, or if BL>ULN then use >2* BL. Urinalysis (Urine protein, urine Glu, urine blood, leukocyte esterase, Red Blood Cells [RBCs], White Blood Cells [WBCs]):Use ≥2 when BL value missing or value ≥4,or when pre-dose=0 or 0.5. Use ≥3 when pre-dose=1. Use ≥4 when pre-dose=2 or 3
Time Frame: Days 1-169
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 428 | 583
participants
  Low Glu (n=427, n=583) | 7 | 17
  High Glu (n=427, n=583) | 12 | 21
  Low protein (n=428, n=583) | 0 | 0
  High protein (n=428, n=583) | 0 | 0
  Low albumin (n=428, n=583) | 1 | 2
  High uric acid (n=428, n=583) | 0 | 0
  High urine protein (n=298, n=421) | 4 | 2
  High urine glucose (n=298, n=421) | 0 | 4
  High urine blood (n=298, n=421) | 5 | 14
  High urine leukocyte esterase (n=297, n=491) | 20 | 17
  High urine RBC (n=68, n=98) | 13 | 17
  High urine WBC (n=80, n=117) | 30 | 36

8. Primary Outcome: Short-term Period: Mean Change From Baseline in Systolic and Diastolic Blood Pressure
Time Frame: Day 1 (Baseline) -Day 169
Population: Although mean values for systolic and diastolic blood pressure were recorded, mean changes from baseline were not summarized for these data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Short-term Period: Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by Enzyme-Linked Immunosorbant Assay (ELISA)
Description: Serum samples from all treated adult participants with active rheumatoid arthritis (RA) were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: Days 1-169
Population: Treated participants with available serum samples for assay
Measure: Number; unit: participants
Groups:
- All Treated Participants: Open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 41
participants
  Anti-abatacept antibodies | 12
  Anti-CTLA4 antibodies | 0

10. Secondary Outcome: Short-term Period: Mean Time-matched Baseline (Day 0) DAS 28 and DAS 28 for Post-Baseline Visits Through 6 Month Open-Label
Description: The DAS 28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: All treated participants. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 429 | 580
units on a scale
  BL (Day 0) for Day 15 cohort (n=429,570) | 6.21 (0.73) | 6.17 (0.72)
  Day 15 visit (n=429,570) | 5.46 (1.05) | 5.49 (1.12)
  BL (Day 0) for Day 29 cohort (n=426,580) | 6.22 (0.72) | 6.17 (0.71)
  Day 29 visit (n=426,580) | 5.05 (1.20) | 5.09 (1.25)
  BL (Day 0) for Day 57 cohort (n=425,563) | 6.22 (0.74) | 6.16 (0.71)
  Day 57 visit (n=425,563) | 4.65 (1.27) | 4.72 (1.30)
  BL (Day 0) for Day 85 cohort (n=403,542) | 6.21 (0.73) | 6.16 (0.72)
  Day 85 visit (n=403,542) | 4.44 (1.37) | 4.57 (1.35)
  BL (Day 0) for Day 113 cohort (n=393,516) | 6.20 (0.73) | 6.15 (0.71)
  Day 113 visit (n=393,516) | 4.24 (1.36) | 4.39 (1.41)
  BL (Day 0) for Day 141 cohort (n=372,493) | 6.19 (0.74) | 6.16 (0.73)
  Day 141 visit (n=372,493) | 4.19 (1.38) | 4.27 (1.39)
  BL (Day 0) for Day 169 cohort(n=369,468) | 6.19 (0.73) | 6.15 (0.73)
  Day 169 visit (n=369,468) | 4.16 (1.43) | 4.14 (1.47)

11. Secondary Outcome: Short-term Period: Mean Time-matched Change From Baseline (Day 0) in DAS 28 Through 6 Month Open-Label
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched mean change from BL= Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL (Day 0) value for only that cohort of participants with measurements available at that post-BL visit.
Time Frame: BL (Day 0), Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: All treated participants. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 429 | 580
units on a scale
  Change from BL (Day 0) to Day 15 visit (n=429,570) | -0.75 (0.04) | -0.68 (0.04)
  Change from BL (Day 0) to Day 29 visit (n=426,580) | -1.18 (0.05) | -1.07 (0.05)
  Change from BL (Day 0) to Day 57 visit (n=425,563) | -1.57 (0.06) | -1.44 (0.05)
  Change from BL (Day 0) to Day 85 visit (n=403,542) | -1.76 (0.06) | -1.60 (0.05)
  Change from BL (Day 0) to Day 113 visit(n=393,516) | -1.96 (0.07) | -1.76 (0.06)
  Change from BL (Day 0) to Day 141 visit(n=372,493) | -2.00 (0.07) | -1.90 (0.06)
  Change from BL (Day 0) to Day 169 visit(n=369,468) | -2.02 (0.07) | -2.01 (0.07)

12. Secondary Outcome: Short-term Period: Mean Change From Baseline to Day 169 in High Sensitivity C-Reactive Protein (Hs-CRP)
Description: hs-CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of hs-CRP can be used to determine DAS28.
Time Frame: BL, Day 169
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 376 | 476
mg/dL | -0.88 (0.13) | -0.68 (0.13)

13. Secondary Outcome: Short-term Period: Mean Change From Baseline to Day 169 in Rheumatoid Factor (RF)
Description: RF is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process.
Time Frame: BL, Day 169
Population: All treated participants
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 376 | 476
IU/mL | -32.2 (11.33) | -22.8 (10.19)

14. Secondary Outcome: Short-term Period: Mean Change From Baseline to Day 169 in the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. HAQ-DI= sum of worst scores in each domain divided by the number of domains answered. HAQ-DI ranges from a minimum of 0 (no difficulty) to a maximum overall score of 3(unable to do).
Time Frame: BL, Day 169
Population: All treated participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 366 | 475
units on a scale | -0.34 (0.03) | -0.41 (0.03)

15. Secondary Outcome: Short-term Period: Number of Participants Achieving a Clinically Meaningful HAQ Response
Description: HAQ-DI includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. HAQ-DI= sum of worst scores in each domain divided by the number of domains answered. HAQ-DI ranges from a minimum of 0 (no difficulty) to a maximum overall score of 3(unable to do). Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ disability Index.
Time Frame: BL, Day 169
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 449 | 597
participants | 208 | 281

16. Secondary Outcome: Short-term Period: Mean Baseline Short Form 36 (SF-36) Quality of Life Physical Component Summary (PCS), Mental Component Summary (MCS), and SF-36 Individual Component Scores
Description: The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: BL
Population: All treated participants. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 370 | 475
units on a scale
  PCS (n=360, n=466) | 28.81 (7.74) | 28.75 (7.47)
  MCS (n=360, n=466) | 42.45 (12.98) | 42.43 (12.43)
  Physical Function Scale Component (n=367, n=473) | 27.72 (9.87) | 28.22 (9.54)
  Role-Physical Scale Component (n=364, n=473) | 32.06 (7.95) | 31.38 (7.11)
  Bodily Pain Scale Component (n=367, n=472) | 31.73 (7.17) | 31.13 (7.26)
  General Health Scale Component (n=369, n=475) | 35.70 (9.40) | 35.71 (9.22)
  Vitality Scale Component (n=369, n=472) | 35.95 (9.21) | 36.62 (9.11)
  Social Functioning Scale Component (n=370, n=475) | 34.76 (11.86) | 34.13 (10.99)
  Role-Emotional Scale Component (n=365, n=471) | 37.21 (13.99) | 36.98 (14.03)
  Mental Health Scale Component (n=369, n=472) | 41.79 (12.79) | 41.92 (11.95)

17. Primary Outcome: Long-term Period: Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuations, AEs, Related AEs, or AEs Leading to Discontinuations
Description: as for outcome 1
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 530
participants
  Death | 1
  SAEs | 61
  Related SAEs | 15
  SAEs Leading to Discontinuation | 11
  AEs | 328
  Related AEs | 146
  AEs Leading to Discontinuation | 15

18. Primary Outcome: Long-term Period: Number of Participants With AEs of Special Interest
Description: as for outcome 2
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 530
participants
  Infections (pre-specified) | 177
  Malignant neoplasms | 4
  Autoimmune disorders (pre-specified) | 8
  Peri-infusional AEs (pre-specified) | 42
  Acute infusional AEs (pre-specified) | 14

19. Primary Outcome: Long-term Period: Number of Participants With Hematology Laboratories Meeting Marked Abnormality (MA) Criteria
Description: ULN=upper limit of normal; LLN=lower limit of normal; BL=baseline. Marked abnormality criteria=Hemoglobin: >3 g/dL decrease from BL; Hematocrit: <0.75*BL; Erythrocytes:<0.75*BL; Platelets: <0.67*LLN/>1.5 * ULN, or if BL<LLN, use 0.5*BL/<100,000 mm^3; Leukocytes: <0.75*LLN/>1.25*ULN, or if BL<LLN, use <0.8*BL/>ULN, or if BL>ULN,use >1.2*BL/<LLN; neutrophils+bands: <1.0*10^3 c/uL; eosinophils: >0.750*10^3 c/uL; basophils: >400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750*10^3 c/uL/>7.50*10^3 c/uL.
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: Participants who received at least 1 infusion of abatacept during the long-term treatment period. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 513
participants
  Low hemoglobin (n=513) | 1
  Low hematocrit (n=510) | 1
  Low erythrocytes (n=513) | 1
  Low platelets (n=500) | 0
  High platelets (n=500) | 1
  Low leukocytes (n=513) | 1
  High leukocytes (n=513) | 8
  Low neutrophils+bands (510) | 0
  Low lymphocytes (n=510) | 34
  High lymphocytes (n=510) | 0
  High monocytes (n=510) | 2
  High basophils (n=510) | 1
  High eosinophils (n=510) | 13

20. Primary Outcome: Long-term Period: Number of Participants With Liver and Kidney Function Laboratories Meeting MA Criteria
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2*ULN, or if BL>ULN, use >3*BL; aspartate aminotransferase (AST): >3*ULN, or if BL>ULN,use >4*BL; alanine aminotransferase (ALT): >3*ULN, or if BL>ULN, use >4*BL; G-Glutamyl transferase (GGT): >2*ULN, or if BL>ULN, use >3*BL; bilirubin: >2*ULN, or if BL>ULN, use >4*BL; blood urea nitrogen (BUN): >2*BL; creatinine: >1.5*BL
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 514
participants
  High ALP (n=514) | 0
  High AST (n=512) | 1
  High ALT (n=512) | 5
  High GGT (n=512) | 10
  High bilirubin (n=513) | 1
  High BUN (n=513) | 5
  High creatinine (n=512) | 8

21. Primary Outcome: Long-term Period: Number of Participants With Electrolyte Laboratories Meeting MA Criteria
Description: as for outcome 6
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 513
participants
  Low Na (n=513) | 1
  High Na (n=513) | 3
  Low K (n=510) | 4
  High K (n=510) | 1
  Low chloride (n=513) | 1
  High chloride (n=513) | 1
  Low Ca (n=513) | 0
  High Ca (n=513) | 1
  Low P (n=512) | 0
  High P (n=512) | 3

22. Primary Outcome: Long-term Period: Number of Participants With Other Chemistry and Urinalysis Laboratories Meeting MA Criteria
Description: as for outcome 7
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable laboratory results.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 513
participants
  Low glu (n=513) | 15
  High glu (n=513) | 17
  Low protein (n=513) | 1
  High protein (n=513) | 0
  Low albumin (n=511) | 1
  High uric acid (n=513) | 0
  High urine protein (n=462) | 4
  High urine glucose (n=462) | 5
  High urine blood (n=462) | 10
  High urine leukocyte esterase (n=462) | 13
  High urine RBC (n=91) | 24
  High urine WBC (n=91) | 11

23. Primary Outcome: Long-term Period: Change From Baseline in Hemoglobin (HGB), Total Protein, and Albumin Over Time
Description: HGB normal range (NR)=11.6 - 16.2 g/dL, marked abnormality (MA) is >3 g/dL decrease from BL. Total protein NR=6.0 - 8.4 g/dL, MA is <0.9* LLN/>1.1* ULN; Albumin NR=3.5 - 5.3 g/dL, MA is <0.9* LLN, or if BL<LLN then use <0.75 BL
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 218
g/dL
  Day 365 HGB (n=218) | 0.40 (0.08)
  Day 365 total protein (n=217) | -0.22 (0.04)
  Day 365 albumin (n=217) | 0.13 (0.02)
  Day 729 HGB (n=62) | 0.47 (0.18)
  Day 729 total protein (n=65) | -0.59 (0.07)
  Day 729 albumin (n=65) | 0.16 (0.04)

24. Primary Outcome: Long-term Period: Change From Baseline in Hematocrit Over Time
Description: The hematocrit value refers to the percentage of blood volume that is occupied by red blood cells. Hematocrit values for participants were expressed as percentages and were averaged to yield a group mean value (percentage) at a particular time point. The mean change from baseline in hematocrit value (expressed as a percent)= mean post-baseline value (expressed as a percent) - mean baseline value (expressed as a percent).
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Long-term ABA
Number analyzed (Participants) | 213
percentage change
  Day 365 hematocrit (n=213) | 1.00 (0.22)
  Day 729 HGB (n=61) | 0.81 (0.47)

25. Primary Outcome: Long-term Period: Change From Baseline in Erythrocytes Over Time
Description: Erythrocytes NR= 3.80 - 5.50 *10^6 c/uL, MA is <0.75 * BL
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: 10^6 c/uL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 218
10^6 c/uL
  Day 365 erythrocytes (n=218) | 0.04 (0.02)
  Day 729 erythrocytes (n=62) | 0.06 (0.04)

26. Primary Outcome: Long-term Period: Change From Baseline in Platelets (PLT) Over Time
Description: Erythrocytes NR= 3.80 - 5.50 *10^6 c/uL, MA is <0.75 * BL
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: 10^9 c/L
Arm/Group | Long-term ABA
Number analyzed (Participants) | 214
10^9 c/L
  Day 365 PLT (n=214) | -41.2 (6.24)
  Day 729 PLT (n=61) | -67.7 (11.02)

27. Primary Outcome: Long-term Period: Change From Baseline in White Blood Cells Over Time
Description: Leukocytes NR=4.1 - 12.3*10^3 c/uL, MA is <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL/>ULN, or if BL>ULN then use >1.2 * BL/<LLN. Neutrophils+bands MA is <1.0 * 10^3 c/uL. Eosinophils MA is >0.750 * 10^3 c/uL. Basophils MA is > 400 mm^3. Monocytes MA is >2000 mm^3. Lymphocytes MA is <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: 10^3 c/uL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 218
10^3 c/uL
  Day 365 leukocytes (n=218) | -0.86 (0.17)
  Day 365 neutrophils (n=215) | -0.83 (0.16)
  Day 365 eosinophils (n=215) | -0.01 (0.01)
  Day 365 monocytes (n=215) | 0.00 (0.02)
  Day 365 basophils (n=215) | 0.00 (0.00)
  Day 365 lymphocytes (n=215) | 0.08 (0.05)
  Day 729 leukocytes (n=62) | -1.49 (0.26)
  Day 729 neutrophils (n=62) | -1.56 (0.27)
  Day 729 eosinophils (n=62) | -0.02 (0.02)
  Day 729 monocytes (n=62) | -0.01 (0.03)
  Day 729 basophils (n=62) | 0.00 (0.00)
  Day 729 lymphocytes (n=62) | 0.10 (0.09)

28. Primary Outcome: Long-term Period: Change From Baseline in Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and G-Glutamyl Transferase (GGT) Over Time
Description: as for outcome 23
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Long-term ABA
Number analyzed (Participants) | 218
U/L
  Day 365 ALP (n=218) | 0.81 (2.64)
  Day 365 AST (n=212) | 0.64 (1.09)
  Day 365 ALT (n=212) | 0.76 (1.80)
  Day 365 GGT (n=217) | 2.21 (3.61)
  Day 729 ALP (n=64) | -8.44 (5.82)
  Day 729 AST (n=63) | 1.35 (2.38)
  Day 729 ALT (n=63) | 2.60 (3.92)
  Day 729 GGT (n=64) | 0.13 (2.34)

29. Primary Outcome: Long-term Period: Change From Baseline in Bilirubin, Blood Urea Nitrogen (BUN), Creatinine, Calcium (Ca), Phosphorus (P), Serum Glucose (Glu), and Uric Acid Over Time
Description: Bilirubin NR=0.2-1.2 mg/dL, MA: >2* ULN, or if BL>ULN then use >4* BL. BUN NR=4.0-24.0 mg/dL, MA: >2*BL. Creatinine NR=0.4-1.2 mg/dL, MA: >1.5*BL. Ca NR=8.8-10.2 mg/dL, MA: <0.8*LLN/>1.2*ULN, or if BL<LLN then use 0.75*BL or >ULN, or if BL>ULN then use>1.25*BL or <LLN. P NR=2.8-4.0 mg/dL, MA: <0.75*LLN/ >1.25*ULN, or if BL<LLN then use 0.67*BL or >ULN, or if BL>ULN then use>1.33*BL or <LLN. Glu MA: <65 mg/dL/ >220 mg/dL. Uric acid MA: >1.5*ULN, or if BL>ULN then use >2*BL.
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 217
mg/dL
  Day 365 bilirubin (n=210) | 0.04 (0.01)
  Day 365 BUN (n=217) | 0.85 (0.31)
  Day 365 creatinine (n=217) | 0.05 (0.01)
  Day 365 Ca (n=217) | 0.11 (0.03)
  Day 365 P (n=217) | 0.13 (0.04)
  Day 365 Glu (n=217) | 0.83 (2.26)
  Day 365 uric acid (n=217) | -0.18 (0.07)
  Day 729 bilirubin (n=65) | -0.01 (0.02)
  Day 729 BUN (n=65) | 0.77 (0.54)
  Day 729 creatinine (n=65) | 0.04 (0.02)
  Day 729 Ca (n=65) | 0.07 (0.06)
  Day 729 P (n=64) | -0.77 (0.08)
  Day 729 Glu (n=64) | 1.71 (2.94)
  Day 729 uric acid (n=65) | 0.11 (0.11)

30. Primary Outcome: LT; Change From Baseline in Sodium (Na), Potassium (K), Chloride (Cl) Over Time
Description: Na NR=132 - 147 mEq/L, MA is 95* LLN/ >1.05* ULN, or if BL<LLN then use 0.95* BL or >ULN, or if BL>ULN then use>1.05* BL or <LLN. K NR=3.3 - 5.5 mEq/L, MA is <0.9* LLN/>1.1* ULN,or if BL<LLN then use 0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN. Cl NR=94 - 111 mEq/L, MA is <0.9* LLN/>1.1* ULN, or if BL<LLN then use 0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN
Time Frame: BL, Day 365, Day 729
Population: All treated participants in the OL. n=number of participants with evaluable laboratory results.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Long-term ABA
Number analyzed (Participants) | 217
mEq/L
  Day 365 Na (n=216) | -0.91 (0.25)
  Day 365 K (n=210) | -0.08 (0.03)
  Day 365 Cl (n=217) | -0.37 (0.25)
  Day 729 Na (n=65) | 1.23 (0.33)
  Day 729 K (n=63) | -0.06 (0.06)
  Day 729 Cl (n=65) | 1.42 (0.37)

31. Primary Outcome: Long-term Period: Mean Sitting Systolic Blood Pressure (SBP) Over Time
Description: Measurements were taken in a seated position before and after abatacept infusion.
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable blood pressure measurements.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Long-term ABA
Number analyzed (Participants) | 482
mm Hg
  Day 169 SBP pre-infusion (n=482) | 125.1 (16.02)
  Day 169 SBP post-infusion (n=478) | 125.3 (16.03)
  Day 197 SBP pre-infusion (n=414) | 124.4 (16.98)
  Day 197 SBP post-infusion (n=415) | 123.9 (16.84)
  Day 225 SBP pre-infusion (n=340) | 123.9 (16.33)
  Day 225 SBP post-infusion (n=338) | 123.4 (16.59)
  Day 253 SBP pre-infusion (n=251) | 124.0 (17.47)
  Day 253 SBP post-infusion (n=251) | 124.9 (16.57)
  Day 281 SBP pre-infusion (n=203) | 124.2 (17.25)
  Day 281 SBP post-infusion (n=202) | 124.8 (16.62)
  Day 309 SBP pre-infusion (n=160) | 124.1 (18.09)
  Day 309 SBP post-infusion (n=159) | 123.8 (17.58)
  Day 337 SBP pre-infusion (n=128) | 124.8 (16.84)
  Day 337 SBP post-infusion (n=128) | 124.0 (18.84)
  Day 365 SBP pre-infusion (n=118) | 126.2 (17.47)
  Day 365 SBP post-infusion (n=120) | 125.0 (15.85)
  Day 393 SBP pre-infusion (n=101) | 123.0 (18.74)
  Day 393 SBP post-infusion (n=99) | 124.1 (17.06)
  Day 421 SBP post-infusion (n=93) | 125.5 (19.44)
  Day 421 SBP post-infusion (n=93) | 124.4 (15.84)
  Day 449 SBP pre-infusion (n=82) | 125.8 (18.29)
  Day 449 SBP post-infusion (n=82) | 124.0 (17.25)
  Day 477 SBP pre-infusion (n=75) | 125.3 (19.03)
  Day 477 SBP post-infusion (n=75) | 122.9 (16.36)
  Day 505 SBP pre-infusion (n=72) | 124.3 (20.88)
  Day 505 SBP post-infusion (n=73) | 122.7 (17.08)
  Day 533 SBP pre-infusion (n=67) | 125.4 (16.73)
  Day 533 SBP post-infusion (n=66) | 125.2 (17.57)
  Day 561 SBP pre-infusion (n=63) | 121.6 (18.36)
  Day 561 SBP post-infusion (n=63) | 120.6 (18.94)
  Day 589 SBP pre-infusion (n=57) | 119.6 (15.98)
  Day 589 SBP post-infusion (n=57) | 121.1 (18.49)
  Day 617 SBP pre-infusion (n=56) | 122.1 (15.62)
  Day 617 SBP post-infusion (n=56) | 122.3 (18.57)
  Day 645 SBP pre-infusion (n=44) | 120.0 (18.78)
  Day 645 SBP post-infusion (n=43) | 121.8 (18.33)
  Day 673 SBP pre-infusion (n=40) | 123.4 (18.53)
  Day 673 SBP post-infusion (n=41) | 123.6 (17.90)
  Day 701 SBP pre-infusion (n=35) | 119.4 (16.82)
  Day 701 SBP post-infusion (n=36) | 117.6 (15.57)
  Day 729 SBP pre-infusion (n=32) | 121.5 (21.43)
  Day 729 SBP post-infusion (n=32) | 121.9 (17.48)
  Day 757 SBP pre-infusion (n=30) | 121.1 (16.36)
  Day 757 SBP post-infusion (n=29) | 118.3 (19.11)
  Day 785 SBP pre-infusion (n=25) | 119.1 (19.97)
  Day 785 SBP post-infusion (n=25) | 117.3 (18.64)
  Day 813 SBP pre-infusion (n=23) | 118.4 (12.24)
  Day 813 SBP post-infusion (n=22) | 123.0 (14.08)
  Day 841 SBP pre-infusion (n=19) | 115.3 (15.92)
  Day 841 SBP post-infusion (n=19) | 119.1 (18.52)
  Day 869 SBP pre-infusion (n=18) | 117.6 (14.84)
  Day 869 SBP post-infusion (n=18) | 117.6 (14.22)
  Day 897 SBP pre-infusion (n=19) | 116.4 (14.18)
  Day 897 SBP post-infusion (n=19) | 115.4 (12.81)
  Day 925 SBP pre-infusion (n=19) | 116.4 (16.33)
  Day 925 SBP post-infusion (n=19) | 118.2 (18.78)
  Day 953 SBP pre-infusion (n=19) | 116.8 (15.97)
  Day 953 SBP post-infusion (n=19) | 119.5 (20.01)
  Day 981 SBP pre-infusion (n=18) | 115.6 (16.18)
  Day 981 SBP post-infusion (n=18) | 118.4 (18.75)
  Day 1009 SBP pre-infusion (n=19) | 116.8 (20.57)
  Day 1009 SBP post-infusion (n=19) | 118.9 (13.70)
  Day 1037 SBP pre-infusion (n=15) | 113.5 (16.51)
  Day 1037 SBP post-infusion (n=15) | 115.3 (15.39)
  Day 1065 SBP pre-infusion (n=14) | 123.1 (24.47)
  Day 1065 SBP post-infusion (n=14) | 119.4 (16.84)
  Day 1093 SBP pre-infusion (n=10) | 116.5 (18.31)
  Day 1093 SBP post-infusion (n=10) | 113.5 (14.54)
  Day 1121 SBP pre-infusion (n=7) | 118.3 (20.93)
  Day 1121 SBP post-infusion (n=7) | 115.1 (11.87)
  Day 1149 SBP pre-infusion (n=7) | 116.9 (13.91)
  Day 1149 SBP post-infusion (n=7) | 116.4 (8.98)
  Day 1177 SBP pre-infusion (n=7) | 114.6 (12.43)
  Day 1177 SBP post-infusion (n=7) | 114.6 (7.72)

32. Primary Outcome: Long-term Period: Mean Sitting Diastolic Blood Pressure (DBP) Over Time
Description: Measurements were taken in a seated position before and after abatacept infusion.
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable blood pressure readings.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Long-term ABA
Number analyzed (Participants) | 481
mm Hg
  Day 169 DBP pre-infusion (n=481) | 75.1 (10.09)
  Day 169 DBP post-infusion (n=477) | 74.9 (9.60)
  Day 197 DBP pre-infusion (n=414) | 74.0 (10.09)
  Day 197 DBP post-infusion (n=415) | 74.4 (10.27)
  Day 225 DBP pre-infusion (n=340) | 73.9 (10.28)
  Day 225 DBP post-infusion (n=338) | 73.7 (9.53)
  Day 253 DBP pre-infusion (n=251) | 74.5 (10.60)
  Day 253 DBP post-infusion (n=251) | 74.5 (10.04)
  Day 281 DBP pre-infusion (n=203) | 74.7 (10.16)
  Day 281 DBP post-infusion (n=202) | 75.3 (9.94)
  Day 309 DBP pre-infusion (n=160) | 75.4 (10.36)
  Day 309 DBP post-infusion (n=159) | 75.6 (10.73)
  Day 337 DBP pre-infusion (n=128) | 74.5 (10.42)
  Day 337 DBP post-infusion (n=128) | 74.5 (10.48)
  Day 365 DBP pre-infusion (n=118) | 76.4 (10.88)
  Day 365 DBP post-infusion (n=120) | 75.0 (10.27)
  Day 393 DBP pre-infusion (n=101) | 75.3 (12.13)
  Day 393 DBP post-infusion (n=99) | 74.7 (10.77)
  Day 421 DBP post-infusion (n=93) | 77.1 (11.66)
  Day 421 DBP post-infusion (n=93) | 75.5 (10.48)
  Day 449 DBP pre-infusion (n=82) | 75.8 (10.82)
  Day 449 DBP post-infusion (n=82) | 76.6 (11.73)
  Day 477 DBP pre-infusion (n=75) | 76.4 (13.25)
  Day 477 DBP post-infusion (n=75) | 75.2 (11.56)
  Day 505 DBP pre-infusion (n=72) | 75.3 (12.80)
  Day 505 DBP post-infusion (n=73) | 75.9 (13.62)
  Day 533 DBP pre-infusion (n=67) | 75.6 (11.36)
  Day 533 DBP post-infusion (n=66) | 77.0 (11.57)
  Day 561 DBP pre-infusion (n=63) | 74.9 (12.10)
  Day 561 DBP post-infusion (n=63) | 73.2 (12.32)
  Day 589 DBP pre-infusion (n=57) | 72.8 (12.0)
  Day 589 DBP post-infusion (n=57) | 74.7 (11.20)
  Day 617 DBP pre-infusion (n=56) | 74.4 (10.92)
  Day 617 DBP post-infusion (n=55) | 74.7 (12.53)
  Day 645 DBP pre-infusion (n=44) | 73.8 (10.68)
  Day 645 DBP post-infusion (n=43) | 76.2 (11.01)
  Day 673 DBP pre-infusion (n=40) | 76.3 (10.32)
  Day 673 DBP post-infusion (n=41) | 75.1 (10.41)
  Day 701 DBP pre-infusion (n=35) | 72.0 (9.39)
  Day 701 DBP post-infusion (n=36) | 72.3 (8.70)
  Day 729 DBP pre-infusion (n=32) | 76.7 (11.66)
  Day 729 DBP post-infusion (n=32) | 74.8 (10.34)
  Day 757 DBP pre-infusion (n=30) | 75.0 (9.34)
  Day 757 DBP post-infusion (n=29) | 73.8 (10.07)
  Day 785 DBP pre-infusion (n=24) | 73.5 (10.46)
  Day 785 DBP post-infusion (n=25) | 72.7 (9.32)
  Day 813 DBP pre-infusion (n=22) | 75.2 (8.05)
  Day 813 DBP post-infusion (n=22) | 73.9 (10.95)
  Day 841 DBP pre-infusion (n=19) | 72.4 (8.41)
  Day 841 DBP post-infusion (n=19) | 73.2 (10.87)
  Day 869 DBP pre-infusion (n=19) | 72.7 (10.61)
  Day 869 DBP post-infusion (n=18) | 71.1 (9.86)
  Day 897 DBP pre-infusion (n=19) | 68.8 (7.44)
  Day 897 DBP post-infusion (n=19) | 67.9 (7.69)
  Day 925 DBP pre-infusion (n=19) | 73.5 (9.96)
  Day 925 DBP post-infusion (n=19) | 71.8 (10.77)
  Day 953 DBP pre-infusion (n=19) | 68.7 (10.91)
  Day 953 DBP post-infusion (n=19) | 72.5 (10.74)
  Day 981 DBP pre-infusion (n=18) | 69.7 (11.05)
  Day 981 DBP post-infusion (n=18) | 69.7 (11.45)
  Day 1009 DBP pre-infusion (n=19) | 71.6 (9.78)
  Day 1009 DBP post-infusion (n=19) | 70.3 (9.16)
  Day 1037 DBP pre-infusion (n=15) | 71.3 (11.15)
  Day 1037 DBP post-infusion (n=15) | 71.2 (8.48)
  Day 1065 DBP pre-infusion (n=13) | 71.5 (7.18)
  Day 1065 DBP post-infusion (n=14) | 72.4 (7.53)
  Day 1093 DBP pre-infusion (n=10) | 71.8 (6.07)
  Day 1093 DBP post-infusion (n=10) | 76.3 (5.58)
  Day 1121 DBP pre-infusion (n=7) | 75.1 (5.64)
  Day 1121 DBP post-infusion (n=7) | 72.6 (4.08)
  Day 1149 DBP pre-infusion (n=7) | 72.6 (4.16)
  Day 1149 DBP post-infusion (n=7) | 72.4 (3.99)
  Day 1177 DBP pre-infusion (n=7) | 69.1 (9.32)
  Day 1177 DBP post-infusion (n=7) | 73.4 (7.35)

33. Primary Outcome: Long-term Period: Mean Heart Rate (HR) Over Time
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable heart rate readings.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Long-term ABA
Number analyzed (Participants) | 481
beats per minute
  Day 169 HR pre-infusion (n=481) | 74.4 (11.08)
  Day 169 HR post-infusion (n=481) | 73.0 (10.22)
  Day 197 HR pre-infusion (n=414) | 74.4 (11.58)
  Day 197 HR post-infusion (n=416) | 72.8 (10.65)
  Day 225 HR pre-infusion (n=340) | 74.7 (10.43)
  Day 225 HR post-infusion (n=338) | 72.5 (9.88)
  Day 253 HR pre-infusion (n=252) | 73.9 (11.72)
  Day 253 HR post-infusion (n=252) | 72.1 (10.96)
  Day 281 HR pre-infusion (n=203) | 73.8 (11.39)
  Day 281 HR post-infusion (n=202) | 72.4 (10.17)
  Day 309 HR pre-infusion (n=160) | 73.9 (9.62)
  Day 309 HR post-infusion (n=159) | 72.0 (9.85)
  Day 337 HR pre-infusion (n=128) | 74.1 (11.71)
  Day 337 HR post-infusion (n=129) | 70.9 (8.78)
  Day 365 HR pre-infusion (n=118) | 73.7 (12.20)
  Day 365 HR post-infusion (n=120) | 73.1 (10.21)
  Day 393 HR pre-infusion (n=101) | 73.0 (10.26)
  Day 393 HR post-infusion (n=99) | 72.4 (9.88)
  Day 421 HR post-infusion (n=93) | 74.2 (10.32)
  Day 421 HR post-infusion (n=93) | 71.6 (8.63)
  Day 449 HR pre-infusion (n=82) | 74.2 (10.67)
  Day 449 HR post-infusion (n=82) | 73.7 (9.81)
  Day 477 HR pre-infusion (n=74) | 75.4 (12.48)
  Day 477 HR post-infusion (n=75) | 72.9 (10.89)
  Day 505 HR pre-infusion (n=72) | 73.8 (11.41)
  Day 505 HR post-infusion (n=73) | 73.0 (8.90)
  Day 533 HR pre-infusion (n=66) | 73.2 (11.57)
  Day 533 HR post-infusion (n=66) | 75.7 (12.21)
  Day 561 HR pre-infusion (n=63) | 73.8 (10.09)
  Day 561 HR post-infusion (n=63) | 72.3 (10.18)
  Day 589 HR pre-infusion (n=57) | 73.0 (9.83)
  Day 589 HR post-infusion (n=57) | 71.5 (9.66)
  Day 617 HR pre-infusion (n=56) | 72.9 (10.89)
  Day 617 HR post-infusion (n=55) | 71.7 (9.40)
  Day 645 HR pre-infusion (n=44) | 76.6 (13.40)
  Day 645 HR post-infusion (n=43) | 76.1 (13.00)
  Day 673 HR pre-infusion (n=40) | 73.5 (11.67)
  Day 673 HR post-infusion (n=41) | 73.3 (10.74)
  Day 701 HR pre-infusion (n=35) | 72.1 (12.13)
  Day 701 HR post-infusion (n=36) | 73.3 (10.23)
  Day 729 HR pre-infusion (n=32) | 70.7 (11.24)
  Day 729 HR post-infusion (n=32) | 71.7 (11.38)
  Day 757 HR pre-infusion (n=30) | 74.1 (9.60)
  Day 757 HR post-infusion (n=30) | 73.2 (9.35)
  Day 785 HR pre-infusion (n=25) | 76.5 (8.78)
  Day 785 HR post-infusion (n=25) | 73.4 (8.61)
  Day 813 HR pre-infusion (n=23) | 73.9 (11.23)
  Day 813 HR post-infusion (n=22) | 71.4 (10.90)
  Day 841 HR pre-infusion (n=19) | 74.2 (10.95)
  Day 841 HR post-infusion (n=19) | 71.4 (9.15)
  Day 869 HR pre-infusion (n=19) | 72.4 (12.21)
  Day 869 HR post-infusion (n=18) | 72.3 (11.98)
  Day 897 HR pre-infusion (n=19) | 71.7 (9.16)
  Day 897 HR post-infusion (n=19) | 70.9 (9.10)
  Day 925 HR pre-infusion (n=19) | 76.7 (7.75)
  Day 925 HR post-infusion (n=19) | 73.0 (7.86)
  Day 953 HR pre-infusion (n=19) | 75.5 (10.57)
  Day 953 HR post-infusion (n=19) | 73.8 (7.49)
  Day 981 HR pre-infusion (n=18) | 75.7 (13.05)
  Day 981 HR post-infusion (n=18) | 72.8 (8.76)
  Day 1009 HR pre-infusion (n=19) | 76.1 (10.68)
  Day 1009 HR post-infusion (n=18) | 73.6 (7.94)
  Day 1037 HR pre-infusion (n=15) | 74.6 (11.36)
  Day 1037 HR post-infusion (n=15) | 75.1 (10.53)
  Day 1065 HR pre-infusion (n=14) | 74.3 (8.90)
  Day 1065 HR post-infusion (n=14) | 75.1 (9.05)
  Day 1093 HR pre-infusion (n=10) | 70.6 (9.54)
  Day 1093 HR post-infusion (n=10) | 70.3 (8.03)
  Day 1121 HR pre-infusion (n=7) | 72.4 (4.89)
  Day 1121 HR post-infusion (n=7) | 69.1 (3.80)
  Day 1149 HR pre-infusion (n=7) | 71.0 (1.83)
  Day 1149 HR post-infusion (n=7) | 69.9 (4.85)
  Day 1177 HR pre-infusion (n=7) | 75.0 (8.85)
  Day 1177 HR post-infusion (n=7) | 69.1 (10.71)

34. Primary Outcome: Long-term Period: Mean Temperature (T) Over Time
Time Frame: From Day 169 through Day 813, including up to 56 days after the last dose of long-term period abatacept
Population: All treated participants. n=number of participants with evaluable temperature readings.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Long-term ABA
Number analyzed (Participants) | 482
degrees Celsius
  Day 169 T pre-infusion (n=482) | 36.5 (0.45)
  Day 169 T post-infusion (n=478) | 36.5 (0.45)
  Day 197 T pre-infusion (n=415) | 36.6 (0.44)
  Day 197 T post-infusion (n=413) | 36.5 (0.43)
  Day 225 T pre-infusion (n=340) | 36.5 (0.48)
  Day 225 T post-infusion (n=335) | 36.5 (0.46)
  Day 253 T pre-infusion (n=251) | 36.5 (0.48)
  Day 253 T post-infusion (n=251) | 36.5 (0.45)
  Day 281 T pre-infusion (n=202) | 36.4 (0.47)
  Day 281 T post-infusion (n=202) | 36.5 (0.45)
  Day 309 T pre-infusion (n=158) | 36.4 (0.48)
  Day 309 T post-infusion (n=158) | 36.4 (0.50)
  Day 337 T pre-infusion (n=129) | 36.3 (0.51)
  Day 337 T post-infusion (n=128) | 36.4 (0.49)
  Day 365 T pre-infusion (n=118) | 36.4 (0.54)
  Day 365 T post-infusion (n=119) | 36.4 (0.55)
  Day 393 T pre-infusion (n=101) | 36.4 (0.47)
  Day 393 T post-infusion (n=96) | 36.4 (0.50)
  Day 421 T post-infusion (n=93) | 36.4 (0.47)
  Day 421 T post-infusion (n=93) | 36.4 (0.45)
  Day 449 T pre-infusion (n=82) | 36.4 (0.44)
  Day 449 T post-infusion (n=82) | 36.4 (0.48)
  Day 477 T pre-infusion (n=75) | 36.4 (0.51)
  Day 477 T post-infusion (n=75) | 36.4 (0.53)
  Day 505 T pre-infusion (n=71) | 36.5 (0.44)
  Day 505 T post-infusion (n=72) | 36.5 (0.55)
  Day 533 T pre-infusion (n=67) | 36.4 (0.57)
  Day 533 T post-infusion (n=64) | 36.4 (0.42)
  Day 561 T pre-infusion (n=63) | 36.4 (0.41)
  Day 561 T post-infusion (n=62) | 36.5 (0.43)
  Day 589 T pre-infusion (n=57) | 36.4 (0.50)
  Day 589 T post-infusion (n=57) | 36.4 (0.47)
  Day 617 T pre-infusion (n=56) | 36.4 (0.51)
  Day 617 T post-infusion (n=54) | 36.4 (0.43)
  Day 645 T pre-infusion (n=44) | 36.3 (0.47)
  Day 645 T post-infusion (n=42) | 36.3 (0.63)
  Day 673 T pre-infusion (n=40) | 36.3 (0.56)
  Day 673 T post-infusion (n=41) | 36.3 (0.50)
  Day 701 T pre-infusion (n=35) | 36.3 (0.49)
  Day 701 T post-infusion (n=35) | 36.3 (0.44)
  Day 729 T pre-infusion (n=31) | 36.1 (0.51)
  Day 729 T post-infusion (n=32) | 36.2 (0.42)
  Day 757 T pre-infusion (n=30) | 36.2 (0.52)
  Day 757 T post-infusion (n=30) | 36.2 (0.53)
  Day 785 T pre-infusion (n=25) | 36.2 (0.40)
  Day 785 T post-infusion (n=24) | 36.2 (0.37)
  Day 813 T pre-infusion (n=23) | 36.1 (0.43)
  Day 813 T post-infusion (n=22) | 36.0 (0.34)
  Day 841 T pre-infusion (n=19) | 36.1 (0.40)
  Day 841 T post-infusion (n=19) | 36.2 (0.46)
  Day 869 T pre-infusion (n=19) | 36.1 (0.66)
  Day 869 T post-infusion (n=18) | 36.1 (0.57)
  Day 897 T pre-infusion (n=18) | 36.2 (0.62)
  Day 897 T post-infusion (n=18) | 36.3 (0.64)
  Day 925 T pre-infusion (n=19) | 36.1 (0.36)
  Day 925 T post-infusion (n=19) | 36.1 (0.43)
  Day 953 T pre-infusion (n=19) | 36.1 (0.54)
  Day 953 T post-infusion (n=18) | 36.1 (0.52)
  Day 981 T pre-infusion (n=17) | 36.2 (0.48)
  Day 981 T post-infusion (n=17) | 36.0 (0.68)
  Day 1009 T pre-infusion (n=19) | 36.1 (0.40)
  Day 1009 T post-infusion (n=17) | 36.3 (0.44)
  Day 1037 T pre-infusion (n=15) | 36.1 (0.38)
  Day 1037 T post-infusion (n=15) | 36.1 (0.41)
  Day 1065 T pre-infusion (n=14) | 36.1 (0.80)
  Day 1065 T post-infusion (n=14) | 36.3 (0.58)
  Day 1093 T pre-infusion (n=10) | 36.1 (0.59)
  Day 1093 T post-infusion (n=10) | 36.2 (0.47)
  Day 1121 T pre-infusion (n=7) | 36.3 (0.40)
  Day 1121 T post-infusion (n=7) | 36.4 (0.33)
  Day 1149 T pre-infusion (n=7) | 36.3 (0.43)
  Day 1149 T post-infusion (n=7) | 36.3 (0.35)
  Day 1177 T pre-infusion (n=7) | 36.1 (0.54)
  Day 1177 T post-infusion (n=7) | 36.2 (0.38)

35. Secondary Outcome: Short-term Period: Mean Change From Baseline to Day 169 in SF-36 PCS, MCS, and SF-36 Individual Component Scores
Description: as for outcome 16
Time Frame: BL, Day 169
Population: All treated participants. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 370 | 475
units on a scale
  PCS (n=360, n=466) | 5.50 (0.44) | 6.08 (0.43)
  MCS (n=360, n=466) | 4.79 (0.59) | 5.43 (0.52)
  Physical Function Scale Component (n=367, n=473) | 4.31 (0.52) | 4.66 (0.49)
  Role-Physical Scale Component (n=364, n=473) | 5.85 (0.59) | 6.82 (0.55)
  Bodily Pain Scale Component (n=367, n=472) | 8.20 (0.45) | 8.72 (0.45)
  General Health Scale Component (n=369, n=475) | 2.85 (0.38) | 3.83 (0.38)
  Vitality Scale Component (n=369, n=472) | 6.32 (0.51) | 6.37 (0.50)
  Social Functioning Scale Component (n=370, n=475) | 6.44 (0.58) | 7.18 (0.54)
  Role-Emotional Scale Component (n=365, n=471) | 5.30 (0.76) | 5.85 (0.71)
  Mental Health Scale Component (n=369, n=472) | 3.74 (0.52) | 4.41 (0.46)

36. Secondary Outcome: Short-term Period: Mean Baseline Fatigue Visual Analog Scale (VAS)
Description: The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on 1 end and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue.
Time Frame: BL
Population: All treated participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 376 | 476
units on a scale | 73.33 (19.67) | 72.70 (20.75)

37. Secondary Outcome: Short-term Period: Mean Change From Baseline to Day 169 in Fatigue Visual Analog Scale (VAS)
Description: as for outcome 36
Time Frame: BL, Day 169
Population: All treated participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ST Abatacept (ABA)-Previous User | ST ABA-Current User
Number analyzed (Participants) | 376 | 476
units on a scale | -18.3 (1.35) | -20.2 (1.25)

38. Secondary Outcome: Long-term Period: Number of Participants With Clinically Meaningful Improvement in DAS 28, Low Disease Activity, or Remission Over Time
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
Time Frame: BL, Days 365, 449, 533, 617, 729, 813
Population: All treated participants. n=number of evaluable participants.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 213
participants
  Day 365 CMI (n=212) | 163
  Day 365 LDAS (n=213) | 70
  Day 365 Remission (n=213) | 31
  Day 449 CMI (n=119) | 105
  Day 449 LDAS (n=120) | 43
  Day 449 Remission (n=120) | 25
  Day 533 CMI (n=102) | 91
  Day 533 LDAS (n=102) | 38
  Day 533 Remission (n=102) | 25
  Day 617 CMI (n=78) | 69
  Day 617 LDAS (n=79) | 38
  Day 617 Remission (79) | 17
  Day 729 CMI (n=59) | 51
  Day 729 LDAS (n=60) | 23
  Day 729 Remission (n=60) | 12
  Day 813 CMI (n=38) | 34
  Day 813 LDAS (n=38) | 21
  Day 813 Remission (n=38) | 12

39. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) DAS 28 and DAS 28 for Post-Baseline Visits Over the Long Term
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched baseline (Day 0)values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: All treated participants analyzed in the LT. N=the total number of participants analyzed, n=the number of participants at that time point with available measurements. Mean time-matched baseline values reflect changing n-values over time
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 212
units on a scale
  BL (Day 0) for Day 365 cohort (n=212) | 6.18 (0.73)
  Day 365 visit (n=212) | 3.90 (1.32)
  BL (Day 0) for Day 449 cohort (n=212) | 6.16 (0.70)
  Day 449 visit (n=212) | 3.55 (1.11)
  BL (Day 0) for Day 533 cohort (n=102) | 6.16 (0.73)
  Day 533 visit (n=102) | 3.52 (1.09)
  BL (Day 0) for Day 617 cohort (n=78) | 6.15 (0.68)
  Day 617 visit (n=78) | 3.44 (1.12)
  BL (Day 0) for Day 729 cohort (n=59) | 6.16 (0.69)
  Day 729 visit (n=59) | 3.49 (1.18)
  BL (Day 0) for Day 813 cohort (n=38) | 6.26 (0.67)
  Day 813 visit (n=38) | 3.28 (1.07)

40. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in DAS 28 Over The Long Term
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched mean change from BL= Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL(Day 0)value for only that cohort of participants with measurements available at that post-BL visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 212
units on a scale
  Change from BL (Day 0) to Day 365 visit (n=212) | -2.28 (0.10)
  Change from BL (Day 0) to Day 449 visit (n=212) | -2.62 (0.11)
  Change from BL (Day 0) to Day 533 visit (n=102) | -2.64 (0.13)
  Change from BL (Day 0) to Day 617 visit (n=78) | -2.72 (0.15)
  Change from BL (Day 0) to Day 729 visit (n=59) | -2.66 (0.19)
  Change from BL (Day 0) to Day 813 visit (n=38) | -2.97 (0.22)

41. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) Number of Tender Joints and Number of Tender Joints for Post-Baseline Visits Over the Long Term
Description: The mean number of tender joints was evaluated based on the number of tender joints in a standard 68 joint count. Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Long-term ABA
Number analyzed (Participants) | 221
tender joints
  BL (Day 0) for Day 365 cohort (n=221) | 16.90 (5.82)
  Day 365 visit (n=221) | 6.04 (6.75)
  BL (Day 0) for Day 449 cohort (n=221) | 16.57 (5.68)
  Day 449 visit (n=221) | 4.39 (5.17)
  BL (Day 0) for Day 533 cohort (n=107) | 16.14 (5.81)
  Day 533 visit (n=107) | 4.34 (4.83)
  BL (Day 0) for Day 617 cohort (n=87) | 16.29 (5.75)
  Day 617 visit (n=87) | 3.75 (4.75)
  BL (Day 0) for Day 729 cohort (n=63) | 16.40 (5.97)
  Day 729 visit (n=63) | 4.02 (5.08)
  BL (Day 0) for Day 813 cohort (n=43) | 17.42 (5.57)
  Day 813 visit (n=43) | 3.67 (4.04)

42. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in Number of Tender Joints Over the Long Term
Description: The mean number of tender joints was evaluated based on the number of tender joints in a standard 68 joint count. Time-matched mean change from baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline (Day 0) value for only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | Long-term ABA
Number analyzed (Participants) | 221
tender joints
  Change from BL (Day 0) to Day 365 visit (n=221) | -10.9 (0.51)
  Change from BL (Day 0) to Day 449 visit (n=221) | -12.2 (0.58)
  Change from BL (Day 0) to Day 533 visit (n=107) | -11.8 (0.70)
  Change from BL (Day 0) to Day 617 visit (n=87) | -12.5 (0.75)
  Change from BL (Day 0) to Day 729 visit (n=63) | -12.4 (0.98)
  Change from BL (Day 0) to Day 813 visit (n=43) | -13.7 (1.12)

43. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) Number of Swollen Joints And Post-Baseline Number of Swollen Joints Over the Long Term
Description: The mean number of swollen joints was evaluated based on the number of swollen joints in a standard 66 joint count. Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Long-term ABA
Number analyzed (Participants) | 221
swollen joints
  BL (Day 0) for Day 365 cohort (n=221) | 12.72 (5.37)
  Day 365 visit (n=221) | 4.56 (4.83)
  BL (Day 0) for Day 449 cohort (n=221) | 12.50 (4.95)
  Day 449 visit (n=221) | 3.63 (3.99)
  BL (Day 0) for Day 533 cohort (n=107) | 11.91 (5.01)
  Day 533 visit (n=107) | 2.81 (2.67)
  BL (Day 0) for Day 617 cohort (n=87) | 11.98 (4.91)
  Day 617 visit (n=87) | 2.97 (3.40)
  BL (Day 0) for Day 729 cohort (n=63) | 11.57 (4.74)
  Day 729 visit (n=63) | 3.02 (4.05)
  BL (Day 0) for Day 813 cohort (n=43) | 12.40 (4.14)
  Day 813 visit (n=43) | 2.14 (3.10)

44. Secondary Outcome: Long-term Period: Mean Time-Matched Change From Baseline (Day 0) in Number of Swollen Joints Over the Long Term
Description: The mean number of swollen joints was evaluated based on the number of swollen joints in a standard 66 joint count. Time-matched mean change from baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline (Day 0) value for only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | Long-term ABA
Number analyzed (Participants) | 221
swollen joints
  Change from BL (Day 0) to Day 365 visit (n=221) | -8.16 (0.40)
  Change from BL (Day 0) to Day 449 visit (n=221) | -8.87 (0.48)
  Change from BL (Day 0) to Day 533 visit (n=107) | -9.09 (0.50)
  Change from BL (Day 0) to Day 617 visit (n=87) | -9.01 (0.60)
  Change from BL (Day 0) to Day 729 visit (n=63) | -8.56 (0.81)
  Change from BL (Day 0) to Day 813 visit (n=43) | -10.3 (0.76)

45. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) Hs-CRP Levels and Hs-CRP Levels for Post-Baseline Over the Long Term
Description: hs-CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of hs-CRP can be used to determine DAS28. Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
mg/dL
  BL (Day 0) for Day 365 cohort (n=216) | 2.36 (2.90)
  Day 365 visit (n=216) | 1.24 (1.78)
  BL (Day 0) for Day 449 cohort (n=125) | 2.48 (2.89)
  Day 449 visit (n=125) | 0.97 (1.59)
  BL (Day 0) for Day 533 cohort (n=106) | 2.65 (2.99)
  Day 533 visit (n=106) | 0.93 (1.39)
  BL (Day 0) for Day 617 cohort (n=80) | 2.82 (3.22)
  Day 617 visit (n=80) | 0.81 (1.21)
  BL (Day 0) for Day 729 cohort (n=61) | 2.47 (3.21)
  Day 729 visit (n=61) | 0.98 (1.57)
  BL (Day 0) for Day 813 cohort (n=43) | 2.60 (2.80)
  Day 813 visit (n=43) | 0.68 (0.96)

46. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in Hs-CRP Level Over the Long Term
Description: hs-CRP is a acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Levels of hs-CRP can be used to determine DAS28. Time-matched mean change from baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline (Day 0) value for only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
mg/dL
  Change from BL (Day 0) to Day 365 visit (n=216) | -1.12 (0.19)
  Change from BL (Day 0) to Day 449 visit (n=125) | -1.51 (0.22)
  Change from BL (Day 0) to Day 533 visit (n=106) | -1.72 (0.26)
  Change from BL (Day 0) to Day 617 visit (n=80) | -2.02 (0.32)
  Change from BL (Day 0) to Day 729 visit (n=61) | -1.49 (0.36)
  Change from BL (Day 0) to Day 813 visit (n=43) | -1.92 (0.43)

47. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) Visual Analog Scale (VAS) and VAS for Post-Baseline Visits Over the Long Term
Description: The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on 1 end and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue. Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit, and represent only that cohort of participants with measurements available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
units on a scale
  BL (Day 0) for Day 365 cohort (n=220) | 74.05 (16.28)
  Day 365 visit (n=220) | 40.61 (24.76)
  BL (Day 0) for Day 449 cohort (n=121) | 73.20 (15.46)
  Day 449 visit (n=121) | 38.74 (24.18)
  BL (Day 0) for Day 533 cohort (n=104) | 73.41 (15.51)
  Day 533 visit (n=104) | 39.27 (23.23)
  BL (Day 0) for Day 617 cohort (n=85) | 73.59 (14.75)
  Day 617 visit (n=85) | 42.16 (22.75)
  BL (Day 0) for Day 729 cohort (n=61) | 73.48 (16.71)
  Day 729 visit (n=61) | 42.90 (23.09)
  BL (Day 0) for Day 813 cohort (n=38) | 74.47 (16.68)
  Day 813 visit (n=38) | 39.61 (22.13)

48. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in VAS Over the Long Term
Description: The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on 1 end and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue. Time-matched mean change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL (Day 0) value for only that cohort of participants with data available at that post-BL visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
units on a scale
  Change from BL (Day 0) to Day 365 visit (n=220) | -33.4 (1.88)
  Change from BL (Day 0) to Day 449 visit (n=121) | -34.5 (2.43)
  Change from BL (Day 0) to Day 533 visit (n=104) | -34.1 (2.82)
  Change from BL (Day 0) to Day 617 visit (n=85) | -31.4 (2.91)
  Change from BL (Day 0) to Day 729 visit (n=61) | -30.6 (3.65)
  Change from BL (Day 0) to Day 813 visit (n=38) | -34.9 (4.03)

49. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) HAQ-DI and HAQ-DI Component Scores For Participant Cohorts at Each Corresponding Post-baseline Visit Over the Long Term
Description: HAQ-DI includes 20 questions to assess physical functions in 8 domains:dressing, arising,eating,walking, hygiene, reach, grip and common activities. Domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. HAQ-DI= sum of worst scores in each domain divided by number of domains answered. HAQ-DI minimum=0 (no difficulty), max overall score=3(unable to do). Time-matched BL(Day 0)values presented for each post-BL visit represent only that cohort of participants with measurements available at that post-BL visit.
Time Frame: BL (Day 0)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
units on a scale
  Day 365 HAQ-DI (n=215) | 1.80 (0.62)
  Day 365 HAQ dressing and grooming (n=215) | 1.62 (0.86)
  Day 365 HAQ arising (n=215) | 1.39 (0.76)
  Day 365 HAQ eating (n=215) | 1.84 (0.92)
  Day 365 HAQ walking (n=215) | 1.43 (0.78)
  Day 365 HAQ hygiene (n=214) | 2.08 (0.77)
  Day 365 HAQ reaching (n=215) | 2.12 (0.80)
  Day 365 HAQ gripping (n=216) | 1.94 (0.70)
  Day 365 HAQ activities (n=216) | 2.00 (0.80)
  Day 449 HAQ-DI (n=116) | 1.89 (0.60)
  Day 449 HAQ dressing and grooming (n=116) | 1.77 (0.81)
  Day 449 HAQ arising (n=116) | 1.45 (0.74)
  Day 449 HAQ eating (n=116) | 2.01 (0.90)
  Day 449 HAQ walking (n=116) | 1.53 (0.76)
  Day 449 HAQ hygiene (n=117) | 2.11 (0.77)
  Day 449 HAQ reaching (n=117) | 2.23 (0.77)
  Day 449 HAQ gripping (n=117) | 1.97 (0.68)
  Day 449 HAQ activities (n=117) | 2.05 (0.76)
  Day 533 HAQ-DI (n=101) | 1.87 (0.62)
  Day 533 HAQ dressing and grooming (n=102) | 1.78 (0.83)
  Day 533 HAQ arising (n=102) | 1.41 (0.76)
  Day 533 HAQ eating (n=102) | 1.96 (0.92)
  Day 533 HAQ walking (n=102) | 1.56 (0.74)
  Day 533 HAQ hygiene (n=101) | 2.07 (0.78)
  Day 533 HAQ reaching (n=101) | 2.22 (0.78)
  Day 533 HAQ gripping (n=101) | 1.96 (0.68)
  Day 533 HAQ activities (n=101) | 2.03 (0.79)
  Day 617 HAQ-DI (n=83) | 1.86 (0.61)
  Day 617 HAQ dressing and grooming (n=83) | 1.78 (0.81)
  Day 617 HAQ arising (n=83) | 1.40 (0.75)
  Day 617 HAQ eating (n=83) | 1.94 (0.90)
  Day 617 HAQ walking (n=83) | 1.54 (0.72)
  Day 617 HAQ hygiene (n=83) | 2.02 (0.76)
  Day 617 HAQ reaching (n=83) | 2.20 (0.78)
  Day 617 HAQ gripping (n=83) | 1.94 (0.69)
  Day 617 HAQ activities (n=83) | 2.04 (0.83)
  Day 729 HAQ-DI (n=63) | 1.86 (0.61)
  Day 729 HAQ dressing and grooming (n=63) | 1.75 (0.82)
  Day 729 HAQ arising (n=63) | 1.40 (0.75)
  Day 729 HAQ eating (n=63) | 1.95 (0.92)
  Day 729 HAQ walking (n=63) | 1.57 (0.67)
  Day 729 HAQ hygiene (n=63) | 2.00 (0.78)
  Day 729 HAQ reaching (n=63) | 2.24 (0.71)
  Day 729 HAQ gripping (n=63) | 1.90 (0.73)
  Day 729 HAQ activities (n=63) | 2.03 (0.80)
  Day 813 HAQ-DI (n=39) | 2.01 (0.62)
  Day 813 HAQ dressing and grooming (n=39) | 1.92 (0.84)
  Day 813 HAQ arising (n=39) | 1.59 (0.75)
  Day 813 HAQ eating (n=39) | 2.18 (0.94)
  Day 813 HAQ walking (n=39) | 1.69 (0.66)
  Day 813 HAQ hygiene (n=39) | 2.10 (0.82)
  Day 813 HAQ reaching (n=39) | 2.41 (0.64)
  Day 813 HAQ gripping (n=39) | 2.00 (0.79)
  Day 813 HAQ activities (n=39) | 2.18 (0.79)

50. Secondary Outcome: Long-term Period: Mean HAQ-DI and HAQ-DI Component Scores For Participant Cohorts at Post-baseline Visits Over the Long Term
Description: HAQ-DI includes 20 questions to assess physical functions in 8 domains:dressing, arising, eating, walking, hygiene, reach, grip and common activities. Domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. HAQ-DI= sum of worst scores in each domain divided by number of domains answered. HAQ-DI minimum=0(no difficulty), max overall score=3(unable to do). Post-BL values presented for each visit represent only that cohort of participants with measurements available at that post-BL visit.
Time Frame: Days 365, 449, 533, 617, 729, 813
Population: All treated participants analyzed in the LT. N=the total number of participants analyzed, n=the number of participants at that time point with available measurements. Mean post-baseline values reflect changing n-values over time
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
units on a scale
  Day 365 HAQ-DI (n=215) | 1.34 (0.75)
  Day 365 HAQ dressing and grooming (n=215) | 1.15 (0.93)
  Day 365 HAQ arising (n=215) | 0.85 (0.80)
  Day 365 HAQ eating (n=215) | 1.26 (1.00)
  Day 365 HAQ walking (n=215) | 1.03 (0.86)
  Day 365 HAQ hygiene (n=214) | 1.70 (1.06)
  Day 365 HAQ reaching (n=215) | 1.73 (1.01)
  Day 365 HAQ gripping (n=216) | 1.45 (0.90)
  Day 365 HAQ activities (n=216) | 1.52 (1.01)
  Day 449 HAQ-DI (n=116) | 1.37 (0.75)
  Day 449 HAQ dressing and grooming (n=116) | 1.17 (0.94)
  Day 449 HAQ arising (n=116) | 0.84 (0.80)
  Day 449 HAQ eating (n=116) | 1.35 (1.03)
  Day 449 HAQ walking (n=116) | 1.02 (0.85)
  Day 449 HAQ hygiene (n=117) | 1.67 (1.02)
  Day 449 HAQ reaching (n=117) | 1.79 (0.96)
  Day 449 HAQ gripping (n=117) | 1.50 (0.91)
  Day 449 HAQ activities (n=117) | 1.61 (1.01)
  Day 533 HAQ-DI (n=101) | 1.33 (0.74)
  Day 533 HAQ dressing and grooming (n=102) | 1.15 (0.95)
  Day 533 HAQ arising (n=102) | 0.82 (0.80)
  Day 533 HAQ eating (n=102) | 1.30 (0.97)
  Day 533 HAQ walking (n=102) | 0.98 (0.87)
  Day 533 HAQ hygiene (n=101) | 1.57 (1.04)
  Day 533 HAQ reaching (n=101) | 1.81 (0.94)
  Day 533 HAQ gripping (n=101) | 1.48 (0.97)
  Day 533 HAQ activities (n=101) | 1.58 (0.94)
  Day 617 HAQ-DI (n=83) | 1.27 (0.68)
  Day 617 HAQ dressing and grooming (n=83) | 0.98 (0.88)
  Day 617 HAQ arising (n=83) | 0.73 (0.81)
  Day 617 HAQ eating (n=83) | 1.33 (0.88)
  Day 617 HAQ walking (n=83) | 0.96 (0.76)
  Day 617 HAQ hygiene (n=83) | 1.48 (0.95)
  Day 617 HAQ reaching (n=83) | 1.70 (0.85)
  Day 617 HAQ gripping (n=83) | 1.43 (0.84)
  Day 617 HAQ activities (n=83) | 1.57 (0.93)
  Day 729 HAQ-DI (n=63) | 1.34 (0.74)
  Day 729 HAQ dressing and grooming (n=63) | 1.03 (0.95)
  Day 729 HAQ arising (n=63) | 0.81 (0.82)
  Day 729 HAQ eating (n=63) | 1.33 (0.97)
  Day 729 HAQ walking (n=63) | 1.11 (0.94)
  Day 729 HAQ hygiene (n=63) | 1.48 (1.03)
  Day 729 HAQ reaching (n=63) | 1.73 (0.81)
  Day 729 HAQ gripping (n=63) | 1.57 (0.91)
  Day 729 HAQ activities (n=63) | 1.68 (0.96)
  Day 813 HAQ-DI (n=39) | 1.38 (0.69)
  Day 813 HAQ dressing and grooming (n=39) | 1.18 (0.97)
  Day 813 HAQ arising (n=39) | 0.82 (0.79)
  Day 813 HAQ eating (n=39) | 1.46 (0.94)
  Day 813 HAQ walking (n=39) | 1.10 (0.79)
  Day 813 HAQ hygiene (n=39) | 1.59 (0.88)
  Day 813 HAQ reaching (n=39) | 1.72 (0.76)
  Day 813 HAQ gripping (n=39) | 1.36 (0.96)
  Day 813 HAQ activities (n=39) | 1.77 (0.93)

51. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in HAQ-DI and HAQ-DI Components For Participant Cohorts at Each Corresponding Post-baseline Visit Over the Long Term
Description: HAQ-DI includes 20 questions assessing physical functions in 8 domains:dressing,arising,eating,walking,hygiene,reach,grip and common activities.Domain questions evaluated on 4-point scale: 0=without any difficulty,1=with some difficulty,2=with much difficulty,and 3=unable to do. HAQ-DI=sum of worst scores in each domain ÷ number of domains answered. HAQ-DI minimum=0 (no difficulty), max overall score=3(unable to do). Time-matched mean change from BL= Post-BL value - time-matched BL value. Time-matched BL value=mean BL (Day 0)value for only that cohort with data available at that post-BL visit.
Time Frame: BL (Day 0), Days 365, 449, 533, 617, 729, 813
Population: as for outcome 39
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Long-term ABA
Number analyzed (Participants) | 216
units on a scale
  Day 365 HAQ-DI (n=215) | -0.46 (0.04)
  Day 365 HAQ dressing and grooming (n=215) | -0.47 (0.06)
  Day 365 HAQ arising (n=215) | -0.54 (0.06)
  Day 365 HAQ eating (n=215) | -0.58 (0.06)
  Day 365 HAQ walking (n=215) | -0.39 (0.05)
  Day 365 HAQ hygiene (n=214) | -0.38 (0.06)
  Day 365 HAQ reaching (n=215) | -0.38 (0.05)
  Day 365 HAQ gripping (n=216) | -0.49 (0.06)
  Day 365 HAQ activities (n=216) | -0.47 (0.06)
  Day 449 HAQ-DI (n=116) | -0.52 (0.05)
  Day 449 HAQ dressing and grooming (n=116) | -0.59 (0.08)
  Day 449 HAQ arising (n=116) | -0.60 (0.07)
  Day 449 HAQ eating (n=116) | -0.66 (0.08)
  Day 449 HAQ walking (n=116) | -0.52 (0.07)
  Day 449 HAQ hygiene (n=117) | -0.44 (0.08)
  Day 449 HAQ reaching (n=117) | -0.44 (0.07)
  Day 449 HAQ gripping (n=117) | -0.47 (0.08)
  Day 449 HAQ activities (n=117) | -0.44 (0.08)
  Day 533 HAQ-DI (n=101) | -0.54 (0.06)
  Day 533 HAQ dressing and grooming (n=102) | -0.64 (0.10)
  Day 533 HAQ arising (n=102) | -0.59 (0.08)
  Day 533 HAQ eating (n=102) | -0.66 (0.10)
  Day 533 HAQ walking (n=102) | -0.58 (0.07)
  Day 533 HAQ hygiene (n=101) | -0.50 (0.09)
  Day 533 HAQ reaching (n=101) | -0.41 (0.09)
  Day 533 HAQ gripping (n=101) | -0.49 (0.10)
  Day 533 HAQ activities (n=101) | -0.45 (0.09)
  Day 617 HAQ-DI (n=83) | -0.59 (0.07)
  Day 617 HAQ dressing and grooming (n=83) | -0.81 (0.10)
  Day 617 HAQ arising (n=83) | -0.66 (0.10)
  Day 617 HAQ eating (n=83) | -0.61 (0.11)
  Day 617 HAQ walking (n=83) | -0.58 (0.09)
  Day 617 HAQ hygiene (n=83) | -0.54 (0.10)
  Day 617 HAQ reaching (n=83) | -0.51 (0.09)
  Day 617 HAQ gripping (n=83) | -0.51 (0.10)
  Day 617 HAQ activities (n=83) | -0.47 (0.10)
  Day 729 HAQ-DI (n=63) | -0.51 (0.09)
  Day 729 HAQ dressing and grooming (n=63) | -0.71 (0.13)
  Day 729 HAQ arising (n=63) | -0.59 (0.12)
  Day 729 HAQ eating (n=63) | -0.62 (0.13)
  Day 729 HAQ walking (n=63) | -0.46 (0.11)
  Day 729 HAQ hygiene (n=63) | -0.52 (0.13)
  Day 729 HAQ reaching (n=63) | -0.51 (0.10)
  Day 729 HAQ gripping (n=63) | -0.33 (0.10)
  Day 729 HAQ activities (n=63) | -0.35 (0.11)
  Day 813 HAQ-DI (n=39) | -0.63 (0.11)
  Day 813 HAQ dressing and grooming (n=39) | -0.74 (0.18)
  Day 813 HAQ arising (n=39) | -0.77 (0.16)
  Day 813 HAQ eating (n=39) | -0.72 (0.18)
  Day 813 HAQ walking (n=39) | -0.59 (0.12)
  Day 813 HAQ hygiene (n=39) | -0.51 (0.17)
  Day 813 HAQ reaching (n=39) | -0.69 (0.13)
  Day 813 HAQ gripping (n=39) | -0.64 (0.14)
  Day 813 HAQ activities (n=39) | -0.41 (0.13)

52. Secondary Outcome: Long-term Period: Number of Participants Achieving Clinically Meaningful HAQ Response Over Time
Description: as for outcome 15
Time Frame: BL, Days 365, 449, 533, 617, 729, 813
Population: All treated participants. N=the total number of participants analyzed, n=the number of participants at that time point with available measurements.
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 215
participants
  Day 365 (n=215) | 124
  Day 449 (n=116) | 69
  Day 533 (n=101) | 62
  Day 617 (n=83) | 53
  Day 729 (n=63) | 38
  Day 813 (n=39) | 26

53. Secondary Outcome: Long-term Period: Mean Time-matched Baseline (Day 0) SF-36 PCS, MCS, and SF-36 Individual Component Scores For Participant Cohorts at Each Corresponding Post-baseline Visit Over the Long Term
Description: SF-36 has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health;(2) mental component summary=vitality,social functioning,role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score and 100=best score. Time-matched BL (Day 0) values presented for each post-BL visit represent only that cohort of participants with measurements available at that post-BL visit
Time Frame: BL (Day 0)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Abatacept (ABA)-Previous User: In participants who had previously used Tumor Necrosis Factor (TNF)-agonists, open-label abatacept was administered on Days 1, 15, and 29 and then once a month thereafter on a background of non-biologic Disease Modifying Anti-Rheumatic Drug (DMARD)s. Participants weighing < 60 kg received 500 mg, participants weighing 60 to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of open-label abatacept by intravenous (IV) infusion.
Arm/Group | Open-label Abatacept (ABA)-Previous User
Number analyzed (Participants) | 306
units on a scale
  Day 365 PCS (n=297) | 28.96 (7.22)
  Day 365 MCS (n=297) | 41.09 (12.90)
  Day 365 Physical Function Scale Component (n=306) | 28.04 (9.88)
  Day 365 Role-Physical Scale Component (n=300) | 31.17 (7.16)
  Day 365 Bodily Pain Scale Component (n=305) | 31.07 (7.39)
  Day 365 General Health Scale Component (n=308) | 35.04 (9.59)
  Day 365 Vitality Scale Component (n=308) | 35.96 (9.11)
  Day 365 Social Functioning Scale Component (n=308) | 34.31 (11.53)
  Day 365 Role-Emotional Scale Component (n=300) | 35.80 (13.80)
  Day 365 Mental Health Scale Component (n=308) | 39.89 (12.86)
  Day 729 PCS (n=83) | 29.76 (6.50)
  Day 729 MCS (n=83) | 36.06 (13.36)
  Day 729 Physical Function Scale Component (n=89) | 26.66 (9.46)
  Day 729 Role-Physical Scale Component (n=85) | 30.87 (6.75)
  Day 729 Bodily Pain Scale Component (n=86) | 29.35 (7.09)
  Day 729 General Health Scale Component (n=90) | 33.23 (9.30)
  Day 729 Vitality Scale Component (n=90) | 36.77 (9.38)
  Day 729 Social Functioning Scale Component (n=90) | 32.59 (12.27)
  Day 729 Role-Emotional Scale Component (n=85) | 30.30 (11.61)
  Day 729 Mental Health Scale Component (n=89) | 33.67 (13.17)

54. Secondary Outcome: Long-term Period: Mean SF-36 PCS, MCS, and SF-36 Individual Component Scores For Participant Cohorts at Each Post-baseline Visits Over the Long Term
Description: SF-36 measures health-related quality of life and has 36 questions with 8 subscale scores and 2 summary scores (1)physical component summary=physical functioning,role-physical,bodily pain,and general health; (2)mental component summary=vitality,social functioning,role-emotional,and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0=worst score and 100=best score. Post-BL values presented for each post-BL visit represent only that cohort of participants with measurements available at that post-BL visit.
Time Frame: Days 365 and 729
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Abatacept (ABA)-Previous User
Number analyzed (Participants) | 306
units on a scale
  Day 365 PCS (n=297) | 35.00 (10.09)
  Day 365 MCS (n=297) | 47.15 (12.80)
  Day 365 Physical Function Scale Component (n=306) | 33.33 (11.45)
  Day 365 Role-Physical Scale Component (n=300) | 37.85 (11.68)
  Day 365 Bodily Pain Scale Component (n=305) | 39.78 (9.87)
  Day 365 General Health Scale Component (n=308) | 38.58 (10.20)
  Day 365 Vitality Scale Component (n=308) | 42.82 (11.27)
  Day 365 Social Functioning Scale Component (n=308) | 41.24 (11.81)
  Day 365 Role-Emotional Scale Component (n=300) | 42.63 (14.32)
  Day 365 Mental Health Scale Component (n=308) | 45.00 (12.82)
  Day 729 PCS (n=83) | 36.92 (9.30)
  Day 729 MCS (n=83) | 42.06 (12.46)
  Day 729 Physical Function Scale Component (n=89) | 33.91 (11.15)
  Day 729 Role-Physical Scale Component (n=85) | 37.61 (11.59)
  Day 729 Bodily Pain Scale Component (n=86) | 38.89 (10.26)
  Day 729 General Health Scale Component (n=90) | 36.99 (9.79)
  Day 729 Vitality Scale Component (n=90) | 42.94 (10.45)
  Day 729 Social Functioning Scale Component (n=90) | 39.28 (11.66)
  Day 729 Role-Emotional Scale Component (n=85) | 37.37 (14.61)
  Day 729 Mental Health Scale Component (n=89) | 40.02 (11.80)

55. Secondary Outcome: Long-term Period: Mean Time-matched Change From Baseline (Day 0) in SF-36 PCS, MCS, and SF-36 Individual Component Scores For Participant Cohorts at Each Corresponding Post-baseline Visit Over the Long Term
Description: SF-36 has 36 questions with 8 subscale scores and 2 summary scores (1)physical component summary=physical functioning,role-physical,bodily pain,and general health; (2)mental component summary=vitality,social functioning,role-emotional,and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0=worst score and 100=best score. Time-matched mean change from BL= Post-BL value - time-matched BL value. Time-matched BL value=mean BL (Day 0)value for only that cohort with data available at that post-baseline visit.
Time Frame: BL (Day 0), Days 365, 729
Population: as for outcome 39
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Open-label Abatacept (ABA)-Previous User
Number analyzed (Participants) | 306
units on a scale
  Day 365 PCS (n=297) | 6.04 (0.55)
  Day 365 MCS (n=297) | 6.06 (0.63)
  Day 365 Physical Function Scale Component (n=306) | 5.29 (0.64)
  Day 365 Role-Physical Scale Component (n=300) | 6.69 (0.68)
  Day 365 Bodily Pain Scale Component (n=305) | 8.70 (0.56)
  Day 365 General Health Scale Component (n=308) | 3.54 (0.46)
  Day 365 Vitality Scale Component (n=308) | 6.86 (0.61)
  Day 365 Social Functioning Scale Component (n=308) | 6.93 (0.67)
  Day 365 Role-Emotional Scale Component (n=300) | 6.83 (0.84)
  Day 365 Mental Health Scale Component (n=308) | 5.11 (0.55)
  Day 729 PCS (n=83) | 7.17 (1.07)
  Day 729 MCS (n=83) | 5.99 (1.27)
  Day 729 Physical Function Scale Component (n=89) | 7.25 (1.31)
  Day 729 Role-Physical Scale Component (n=85) | 6.74 (1.25)
  Day 729 Bodily Pain Scale Component (n=86) | 9.54 (1.12)
  Day 729 General Health Scale Component (n=90) | 3.76 (0.99)
  Day 729 Vitality Scale Component (n=90) | 6.16 (1.09)
  Day 729 Social Functioning Scale Component (n=90) | 6.69 (1.47)
  Day 729 Role-Emotional Scale Component (n=85) | 7.06 (1.50)
  Day 729 Mental Health Scale Component (n=89) | 6.35 (1.16)

56. Secondary Outcome: LT; Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by ELISA
Description: as for outcome 9
Time Frame: Days 1-813
Population: Treated participants with available serum samples for assay
Measure: Number; unit: participants
Arm/Group | Long-term ABA
Number analyzed (Participants) | 25
participants
  Anti-abatacept antibodies | 0
  Anti-CTLA4 antibodies | 0

ADVERSE EVENTS:
Arm/Group | Abatacept (LT) | Abatacept (ST)
Serious Adverse Events (participants affected / at risk) | 61/530 | 110/1046
Other Adverse Events (participants affected / at risk) | 130/530 | 372/1046
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (LT) (N=530) | Abatacept (ST) (N=1046)
MEDICAL OBSERVATION (Investigations) | 0 | 2
BLOOD SODIUM DECREASED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1
CARDIOMEGALY (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
SINOATRIAL BLOCK (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 3
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 0
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
SHOCK (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 1
AORTIC STENOSIS (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
SUICIDAL BEHAVIOUR (Psychiatric disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1
GALLBLADDER ENLARGEMENT (Hepatobiliary disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 1
SCIATICA (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
CERVICAL ROOT PAIN (Nervous system disorders) | 1 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 2
COLITIS (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 1 | 0
RETCHING (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
PROCTITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 4
UROSEPSIS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 3
BACTERAEMIA (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 1
ACUTE SINUSITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 3 | 1
LOBAR PNEUMONIA (Infections and infestations) | 0 | 2
TOOTH INFECTION (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 1
ABSCESS INTESTINAL (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 1
HAEMOPHILUS INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 | 1
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 2
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
MESANGIOPROLIFERATIVE GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 1
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1
POLYMENORRHOEA (Reproductive system and breast disorders) | 0 | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 | 5
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 15 | 17
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 3
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY BULLA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ULCER (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 3 | 4
CHEST DISCOMFORT (General disorders) | 0 | 2
IMPAIRED HEALING (General disorders) | 0 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (LT) (N=530) | Abatacept (ST) (N=1046)
HEADACHE (Nervous system disorders) | 25 | 102
NAUSEA (Gastrointestinal disorders) | 26 | 90
DIARRHOEA (Gastrointestinal disorders) | 24 | 58
SINUSITIS (Infections and infestations) | 24 | 63
BRONCHITIS (Infections and infestations) | 30 | 49
NASOPHARYNGITIS (Infections and infestations) | 34 | 32
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 25 | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.